CLINICAL TRIAL: NCT07124338
Title: Preventing Hospital Associated Disability in Older Patients: Individualized Nutrition and Exercise Strategy, a Feasibility Study
Acronym: PrevHAD FS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Charlotte Suetta, Professor, Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: p-2025-18713; 3165-00244B (Other Grant/Funding Number: Independent Research Fund Denmark)
Record Dates: First submitted 2025-07-03; First posted 2025-08-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenia in Elderly; Hospital Associated Deconditioning; Malnutrition Elderly; Physical Function
Keywords: Older; Hospitalized; hospital associated disability; Sarcopenia; Malnutrition; Nutritional intervention; Exercise intervention
MeSH Terms: conditions — Sarcopenia; Malnutrition | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Feasibility Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise and nutrition intrvention (Experimental): During hospitalization, 2x 30 minutes of supervised exercise. Furthermore during hospitalization, an inital nutrition plan by a trained dietician, based on Nutrional risk, identifying of nutrion impact symtomes, daily nutritional intake regristration and adjustments to the nutrion plan
  Interventions: Other: Exercise, supervised

INTERVENTIONS:
Other: Exercise, supervised — nital nutrition plan by a trained dietician, based on Nutritional risk, identifying of nutrion impact symtomes, daily nutritional intake regristration and adjustments to the nutrion plan

SUMMARY:
Aproximately a third of persons older than 70 years lose physical function and ability to take care of themselves during a stay at a hospital. This is associated to an increased risk of readmission and mortality. Earlier research has shown that insufficient nutrition and physical activity during hospital stay, leading to a loss in muscle mass and strength, plays an important role in this fall in functionality. This study aims to examine if a structured and supervised resistance exercise, with or without an individualized nutritional plan and intervention, can prevent this fall in functional ability during hospital stay among older patients.

Furthermore, this study seeks to investigate if it is feasible to carry out such a exercise and nutritional intervention in a hospital setting, and to obtain viewpoints regarding exercise and nutrition during hospital stay from older patients. This study aims to produce experience for at bigger randomized controlled study expected later in 2025

DETAILED DESCRIPTION:
Introduction Older persons are highly susceptible to hospital associated disability (HAD), defined by a loss of physical function during hospitalization, leading to increased dependency, morbidity, and mortality. Key factors in developing HAD are physical inactivity, malnutrition and dehydration, leading to a decline in muscle mass and muscle strength. Therefore, there is a need to develop effective nutritional and exercise interventions for older patients, during hospitalization.

Hypothesis This study expects that a mobility-graded individualized exercise intervention will effectively prevent a decline in activities of daily living (ADL) function, mobility level, physical function, muscle and strength, and reduce the length of stay, risk of re-admission and mortality among older patients during hospital stay. The investigators furthermore hypothesize that the combined effect of exercise and optimized nutrition/hydration will be more effective compared to exercise and standard care, and additionally improve the nutritional and hydrational status and lower risk of delirium during hospital stay.

Before initiating a large scale RCT, a study examining the feasibility of the design will be performed.

The Feasibility-pilot study will include 25 participants, men and women, ≥ 65 years old from the geriatric care unit of Bispebjerg Hospital, Denmark. After inclusion, participants will have estimated nutritional status, frailty and mobility, muscle mass and strength, physical function, ADL function and quality of life. The Participants will receive 2 x 30 supervised exercis and a personalized nutritional plan, including refeeding risk management. In addition, the participants will be interviewed approximately 20 minutes the day before discharge. Based on predefined progression criteria using the traffic light model and qualitative feedback from the participants obtained from interviews and a new power calculation of sample size based on representative baseline characteristics, changes to design in the following RCT will be made.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at the geriatric ward
* Speak Danish or English
* Ability to give informed consent

Exclusion Criteria:

* Moderate to severe Dementia¨
* Manifest delirium
* Requiring specialized diet (allergies, diseases requiring special diets, aiming to lose weight)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Eligibility to enter the study | on inclusion day
  75 % or more of screened patients eligible to enter the study, based on exclusion and inclusion criteria.

SECONDARY OUTCOMES:
Inclusion and recruitment | on inclusion day
  1 participant included pr weekday and more than 75% of eligible patients accept inclusion after proposal
Adherence to protocol: Exercise team workflow | From inclusion to discharge from the geriatric department, varying fror each participant, but estimated 3-14 days.
  90 % of planned exercise bouts initiated.
Adherence to protocol: Exercise outcome | From inclusion to discharge from the geriatric department, varying fror each participant, but estimated 3-14 days.
  85 % of initiated exercise bouts completed with 75 % of planned exercise
Adherence to protocol: Dietician workflow | Inclusion day
  95 % or more of participants in nutrition intervention group receiving an individualized nutritional plan on inclusion day
Adherence to protocol: Nutrition outcome | Four days after inclusion
  80 % of participants with 75 % or more of planned daily caloric intake 4 days after admission
Outcome data: Barthel index 100 | At inclusion and again at discharge from the geriatric department, varying for each participant, but estimated 3-14 days after inclusion.
  90 % of included participants with data collection on planned RCT substudy 1 primary outcomes (Barthel Index 100 (0-100, 0 complete dependency in ADL function, 100 complete independence in ADL function)
Outcome data: Secondary (Cumulated Ambulation Score) | At inclusion and again at discharge from the geriatric department, varying for each participant, but estimated 3-14 days after inclusion.
  75 % of included participants with data collection on planned RCT secondary outcomes Cumulated Ambulation Score (assesed mobility, 0-6)
Adverse effects | From inclusion to discharge from the geriatric department, varying fror each participant, but estimated 3-14 days.
  No falls or function-limiting injuries related to exercise, few minor injuries. No cases of manifest refeeding syndrome related to the nutrition intervention.
Assessment duration | At inclusion and again at discharge from the geriatric department, varying for each participant, but estimated 3-14 days after inclusion.
  All assessments completed faster than 120 minutes
Dropout | From inclusion to discharge from the geriatric department, varying fror each participant, but estimated 3-14 days.
  Less than 15 % dropout of included participants
Outcome data: Primary, Knee extension strength | At inclusion and again at discharge from the geriatric department, varying for each participant, but estimated 3-14 days after inclusion.
  90 % of included participants with data collection on planned RCT substudy 2 primary outcomes (Knee extension strength, maximal voluntary contraction, newton meter)
Outcome data: Secondary (Hand grip strength ) | At inclusion and again at discharge from the geriatric department, varying for each participant, but estimated 3-14 days after inclusion.
  75 % of included participants with data collection on planned RCT secondary outcomes: Hand grip strength, kilogram
Outcome data: Secondary (Sit-to-stand test ) | At inclusion and again at discharge from the geriatric department, varying for each participant, but estimated 3-14 days after inclusion.
  75 % of included participants with data collection on planned RCT secondary outcomes: Sit-to-stand test, number of repetitions in 30 seconds, continous scale
Outcome data: Secondary (Gait speed) | At inclusion and again at discharge from the geriatric department, varying for each participant, but estimated 3-14 days after inclusion.
  75 % of included participants with data collection on planned RCT secondary outcomes: Gait speed, velocity (meters/seconds)
Outcome data: Secondary (Quadriceps muscle thickness) | At inclusion and again at discharge from the geriatric department, varying for each participant, but estimated 3-14 days after inclusion.
  75 % of included participants with data collection on planned RCT secondary outcomes: Quadriceps muscle thickness, ultrasound, millimeters
Outcome data: Secondary (muscle mass) | At inclusion and again at discharge from the geriatric department, varying for each participant, but estimated 3-14 days after inclusion.
  75 % of included participants with data collection on planned RCT secondary outcomes: muscle mass, bioimpedance analysis, kilogram
Outcome data: Secondary (appetite) | At inclusion and again at discharge from the geriatric department, varying for each participant, but estimated 3-14 days after inclusion.
  75 % of included participants with data collection on planned RCT secondary outcomes: appetite, simplified nutritional appettite questionaire.
Outcome data: Secondary (quality of life) | At inclusion and again at discharge from the geriatric department, varying for each participant, but estimated 3-14 days after inclusion.
  75 % of included participants with data collection on planned RCT secondary outcomes: quality of life, EuroQol- 5D-5 levels questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Suetta, Professor, Principal Investigator — Geriatric research unit, Bispebjerg hospital, Copenhagen
Locations (1):
- Bispebjerg Hospital, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
We will share the protocol for the exercise and nutrional intervention, As well as participants charecteristics and outcome data, in a data repository, when the data can be fully anonymized
Access Criteria: Data repository, URL link within the published feasibility study